CLINICAL TRIAL: NCT04658043
Title: Early Socioemotional Intervention for Children With Autism Spectrum Disorder in Hong Kong and Mainland China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Shenzhen University (Other); Guangdong Province, Department of Science and Technology (Other Government)
Responsible Party: Principal Investigator, Professor Terry Kit-fong Au, Vice-President and Pro-Vice-Chancellor (Academic Staffing and Resources), The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EA1811014
Record Dates: First submitted 2020-11-10; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; ASD; socioemotional functioning; Intervention study
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD Intervention Group (Experimental): Participants in the ASD intervention group will receive training to help children improve socioemotional functioning.
  Interventions: Other: Intervention on socioemotional functioning
- Wait List Control Group (No Intervention): Participants in this group will be placed on the wait list and receive the ASD intervention training 2 months after the other groups

INTERVENTIONS:
Other: Intervention on socioemotional functioning — A culturally sensitive intervention based on the "train the trainer (or coach the coach) model" for enhancing the social adaptive functioning of young children (aged 3-6) with ASD in China, via providing training for parents
  Arms: ASD Intervention Group

SUMMARY:
This study aims to develop a culturally-sensitive parent-training intervention to enhance socioemotional functioning of young children (aged 3-6) with Autism Spectrum Disorder (ASD) in Mainland China. The investigators will conduct randomized controlled trials to evaluate the effectiveness and feasibility of this program in a pilot study and then a large-scale community-based study in Shenzhen, China, to examine the generalizability of the treatment outcomes of this intervention for Chinese children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-6
* Living in Shenzhen, Mainland China
* Diagnosed with ASD or suspected of having ASD

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-22 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) | pre-intervention and 4-month post-intervention
  ADOS-2 is a diagnostic measure used in this study to assess the change in children's ASD symptoms
Change in the Autism Spectrum Quotient (AQ) | pre-intervention, immediately after the intervention, and 4-month post-intervention
  AQ is a parent-report measure used in this study to measure change in children's ASD symptoms
Change in Dyadic Parent-Child Interaction Coding System (DPICS system) | pre-intervention, immediately after the intervention, and 4-month post-intervention
  The DPICS system is used in this study to measure the change in the quality of parent-child interaction through observations of dyads during free and structured play in the clinical setting and 5-minute parents' description of their children. The code categories include the number of command, praise, joint attention and verbal responsiveness, words used by parents and the intonation in their language.

SECONDARY OUTCOMES:
Change in Parenting Stress Index, Fourth Edition Short Form (PSI-4-SF) | pre-intervention, immediately after the intervention, and 4-month post-intervention
  PSI-4-SF is a parent-report measure used in this study to measure change in parenting stress
Change in Self-Efficacy in Nurturing Role Questionnaire | pre-intervention, immediately after the intervention, and 4-month post-intervention
  Self-Efficacy in Nurturing Role Questionnaire is a parent-report measure used in this study to measure change in parents' self-efficacy
Change in Classroom Observation Scale (COS) | pre-intervention, immediately after the intervention, and 4-month post-intervention
  COS is a teacher-report measure used in this study to measure children's social behaviours in classroom setting
Change in Social Responsiveness Scale, Second Edition (SRS-2) | pre-intervention, immediately after the intervention, and 4-month post-intervention
  SRS-2 is a teacher-report measure used in this study to measure children's social behaviours

CONTACTS AND LOCATIONS:
Overall Officials: Terry Kit-fong Au, Principal Investigator — The University of Hong Kong
Locations (2):
- Shenzhen University, Shenzhen, China
- University of Hong Kong, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Informed Consent Form (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04658043/ICF_000.pdf